CLINICAL TRIAL: NCT02091011
Title: LONGEVITY Study. Evaluation of the Device and Battery Longevity of Boston Scientific Market-released ICD and CRT-D Devices.
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PDM 90912475
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Implantable Cardioverter Defibrillators; CRT-D Cardiac Resynchronization Therapy Defibrillator
Keywords: This study is designed to efficiently provide device and battery longevity data on market released; Boston Scientific ICD and CRT-D (Cardiac Resynchronization Therapy Defibrillator) devices. In addition, the data collected will allow for; comparisons of device survival probability estimated in the Product Performance Report versus; those collected in the study. The data collected will also provide a better understanding on the; potential predictors of pulse generator battery longevity.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort group: Subjects who have been implanted within 30 days with a commercially available Boston Scientific ICD or a CRT-D device

SUMMARY:
The study is to determine the rate and cause of device replacements at 5 years post-implantation. It will assess the battery and device longevity of the Implantable Cardioverter Defibrillators (ICD) and CRT-D Cardiac Resynchronization Therapy Defibrillator (CRT-D) devices. It will also validate the device survival information given in Boston Scientific's Product Performance Report by comparing the pulse generator (PG) survival probability in the study to that presented in the Product Performance Reports (PPR)

ELIGIBILITY:
Inclusion Criteria:

* Subject has been implanted within 30 days with a commercially available Boston Scientific ICD or a CRT-D device according to current guidelines and/or center's current practice
* Subject is willing and capable (or appropriate legal representative is willing and capable) of authorizing access to and use of health information as required by an Institution's Institutional Review Board (IRB), Research Ethics Board (REB) or Ethics Committee (EC)
* Is willing and capable (or appropriate legal representative is willing and capable) of providing authorization/consent for participation in the study.

Exclusion Criteria:

* Subject is unable or unwilling to comply with the study protocol requirements
* Subject is under the legal age for signing study consent in accordance with state or national law
* Subject has a life expectancy of less than twelve months
* Women of childbearing potential who are or might be pregnant at the time of study enrollment (method of assessment upon physician's discretion)
* Subject on active heart transplant list
* Subject with any prior pulse generator infection or lead infection which is either systemic or localized
* Subject received a commercially available Boston Scientific ICD or CRT-D device with a battery capacity of 1.5 amp/hour or less
* Subject implanted with Boston Scientific's subcutaneous implantable defibrillator system (s-ICD) or has a lead that is under recall/advisory at the time of enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject has been implanted within 30 days with a commercially available Boston Scientific ICD or a CRT-D device according to current guidelines and/or center's current practice
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Determine the rate and cause of all-cause device replacements of Boston Scientific's market-released ICD and CRT-D devices at 5 years post-implantation. | 5 years
Evaluate the battery survival of Boston Scientific's market-released ICD and CRT-D devices at 5 years post-implantation. | 5 years
  Battery survival is defined as freedom from surgical replacement of the device due to battery depletion.

SECONDARY OUTCOMES:
Determine the rate and cause of all-cause device replacement of Boston Scientific's market-released ICD and CRT-D devices 1, 2, 3 and 4 years post-implantation. | 1, 2, 3, and 4 years
Evaluate battery survival of Boston Scientific's market-released ICD and CRT-D devices at 1, 2, 3 and 4 years post-implantation. | 1, 2, 3, and 4 years
Evaluate the device survival of Boston Scientific's market released ICD and CRT-D pulse generators at 5 years post-implantation; and compare it to the survival probability presented in the Product Performance Report (PPR). | 5 years
Evaluate potential predictors of device battery longevity at 5 years post-implantation. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Samir Saba, MD, FACC, FHRS, Principal Investigator — University of Pittsburgh Medical Center
Locations (80):
- United States (51):
  - Alabama cardiovascular group, Birmingham, Alabama
  - Birmingham Heart Clinic, P.C., Birmingham, Alabama
  - Phoenix Heart, PLLC, Glendale, Arizona
  - Pima Heart Physicians PC, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Mercy Clinic Cardiology Physician Plaza, Rogers, Arkansas
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Bradenton Cardiology Center, Bradenton, Florida
  - Jackson Memorial Hospital, JHS Office of Research, Miami, Florida
  - Florida Electrophysiology, LLC, Orlando, Florida
  - Bay Area Heart Center, St. Petersburg, Florida
  - Alexian Brothers, Elk Grove Village, Illinois
  - Franciscan Physician Network Cardiology Crown Point, Crown Point, Indiana
  - The Heart Group, PC, Newburgh, Indiana
  - InityPoint Health - St. Luke's Hospital, Cedar Rapids, Iowa
  - Advance Cardiovascular Specialists, Shreveport, Louisiana
  - Delmarva Heart Research Foundation, Inc., TidalHealth Peninsula Regional, Inc., Salisbury, Maryland
  - Mass Heart and Rhythm, Leominster, Massachusetts
  - McLaren Bay, Bay City, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Great Lakes Heart And Vascular Institute, Saint Joseph, Michigan
  - Cardiovascular Clinic of Hattiesburg, Hattiesburg, Mississippi
  - Wesley Medical Center, Hattiesburg, Mississippi
  - Kansas City Heart Foundation, Kansas City, Missouri
  - PCRMC Medical Group, Rolla, Missouri
  - Gateway Cardiology, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - University Hospital, Newark, Newark, New Jersey
  - Stony Brook Community Medical, PC, East Setauket, New York
  - New York Hospital Queens, Flushing, New York
  - Westchester Heart & Vascular, Hawthorne, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Stark Medical Specialties, Massillon, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Cardiology Sacred Heart at Riverbend Hospital, Springfield, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Heart and Vascular Institute, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Carolina Cardiology Assoc, Piedmont Medical Center, Rock Hill, South Carolina
  - Parkridge Medical Ctr., Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Heart Rhythm, Houston, Texas
  - Cardiology Clinic San Antonio, San Antonio, Texas
  - Central Utah Clinic, Provo, Utah
  - Cardiology Associates of Fredericksburg, Fredericksburg, Virginia
  - Carient Heart & Vasculare, Manassas, Virginia
  - CAMC Health Education and Research Institute, Charleston, West Virginia
  - Prevea Clinic, Inc., Green Bay, Wisconsin
  - Clinical Research Specialist, Research Institute ProHealth Care, Inc, Waukesha, Wisconsin
- Canada (4):
  - Cardiology Research Group Royal Alexandra Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Hospital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, CHUS/CRC, Sherbrooke, Quebec
- Germany (2):
  - Charite Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Schleswig-Holstein, Klinik für Kardiologie und Angiologie, Kiel
- Japan (7):
  - Chiba University Hospital, Chiba
  - Fukuoka University Hospital, Fukuoka
  - University of Tsukuba Hospital, Ibaraki
  - Japan Labour Health and and Welfare Organization, Yokohama Rosai Hospital, Kanagawa-Prefecture
  - Saitama Medical University, Saitama Redcross Hospital, Saitama
  - Tokohu University Hospital, Sendai
  - Showa University Hospital, Tokyo
- South Korea (7):
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary Hospital, Seoul
  - Sejong General Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul
- Spain (3):
  - Hospital Universitario de Cruces. Servicio de Cardiología, Barakaldo
  - Hospital Universitario La Paz. Servicio de Cardiología. Sección de Arritmias. Planta primera diagonal, Madrid
  - Hospital Universitario "Miguel Servet". Servicio de Cardiología, Zaragoza
- Switzerland (2):
  - Universitatsspital Basel Klinik fur Kardiologie, Basel
  - Kantonspital St Gallen, Klinik fur Kardiologie, Sankt Gallen
- United Kingdom (4):
  - Bristol Heart Institute, Bristol
  - St Bartholomew's Hospital, EP Cardiac Research Department, Barts Health NHS Trust, London
  - James Cook University Hospital, Middlesbrough
  - University Hospital of Southhampton, Southampton